CLINICAL TRIAL: NCT03043508
Title: Overall and Disease Specific Survival in Patients With Confirmed MEN1 With or Without PNET (Pancreatic Neuroendocrine Tumors)
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA15-0231
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Genetic Mutation; MEN1
Keywords: Genetic mutation; MEN1; Pancreatic neuroendocrine tumor; PNET; Chart review; Questionnaire; Survey
MeSH Terms: conditions — Adenoma, Islet Cell; Neuroectodermal Tumors, Primitive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants With Confirmed MEN1 With PNET: Retrospective review of a prospectively maintained MEN1 database.
  Participants sent an email questionnaire to complete regarding their pregnancy and hormone use history.
  Interventions: Other: Chart Review; Behavioral: Questionnaire
- Participants With Confirmed MEN1 Without PNET: Retrospective review of a prospectively maintained MEN1 database.
  Participants sent an email questionnaire to complete regarding their pregnancy and hormone use history.
  Interventions: Other: Chart Review; Behavioral: Questionnaire

INTERVENTIONS:
Other: Chart Review — Database reviewed to obtain patient and disease characteristics, laboratory values, imaging results, hormone parameters (menopausal status, bioidentical hormone use, oral contraception use, gestational status and diagnosis of a prolactinoma) and vital status.
Behavioral: Questionnaire — Participants sent an email questionnaire to complete regarding their pregnancy and hormone use history.
  Other Names: Survey

SUMMARY:
OBJECTIVES:

The primary objective of this study is to evaluate the effect of estrogen on the development of the PNET in MEN1 patients.

The secondary objective is to evaluate the overall survival and disease specific survival in patients who have confirmed MEN1 with or without PNET and a pancreatic neuroendocrine tumor in relation to their hormone status. The secondary objective is to evaluate clinicopathologic features in relation to hormone status.

DETAILED DESCRIPTION:
Retrospective review of a prospectively maintained MEN1 database. The patient cohort consists of all patients with confirmed MEN1 with or without PNET who are included in the database. The database will be reviewed to obtain patient and disease characteristics, laboratory values, imaging results, hormone parameters (menopausal status, bioidentical hormone use, oral contraception use, gestational status and diagnosis of a prolactinoma) and vital status.

For the prospective portion of this study, investigators want to see the impact of estrogen on the PNET forming and progression, and would like to use two equations to assess the estrogen exposure, so investigators should collect the information of menopause, menarche, breast feed, HRT, OCP use and pregnancy. To this end, investigators will contact female patients in the database who are still living, and obtain verbal informed consent to send an email questionnaire regarding their pregnancy and hormone use history.

ELIGIBILITY:
Inclusion Criteria:

1. The patient cohort for this study consists of all patients within the prospectively maintained MEN1 database within the Department of Surgical Oncology at the University of Texas MD Anderson Cancer Center.
2. Patients with a diagnosis of MEN1 with or without PNET based on mutational analysis or defined clinical criteria were considered.
3. All patients for whom hormone status variables and survival data are available will be included.

Exclusion Criteria:

1. Due to the nature of the questions included in the prospective estrogen questionnaire, only female patients will be verbally consented to receive the questionnaire and obtain prospective data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Prospectively maintained MEN1 database within the Department of Surgical Oncology, Division of Surgical Endocrinology at the University of Texas MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to Pancreatic Neuroendocrine Tumors (PNET) | 10 years
  Time to PNET calculated starting from the date of menarche time to the PNET diagnostic date or the menopause date (for the patients who get the menopause prior to the PNET diagnosis) or the last follow-up date.

SECONDARY OUTCOMES:
Overall Survival in Participants Who Have Confirmed MEN1 with or without PNET | 10 years
  Overall survival estimated and plotted using Kaplan-Meier method (Kaplan, 1958)(4).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org